CLINICAL TRIAL: NCT01635452
Title: A Prospective Multicenter Non-interventional Study of Women Treated With ESMYA (Ulipristal Acetate) as Pre-operative Treatment of Moderate to Severe Symptoms of Uterine Fibroids
Acronym: PREMYA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: PregLem SA (Industry)
Responsible Party: Sponsor
Other Study IDs: PGL10-014
Record Dates: First submitted 2012-06-26; First posted 2012-07-09 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients treated with Esmya

SUMMARY:
This is a multi-center, prospective, non-interventional study of patients who have been diagnosed with moderate to severe symptoms of uterine fibroids and are initiating a pre-operative treatment with ESMYA.

The objectives of the study are to characterize and describe treatment with ESMYA and to evaluate the safety, effectiveness, and HRQL outcomes in this population

ELIGIBILITY:
Inclusion Criteria:

- Pre-menopausal adult women with a diagnosis of moderate or severe symptoms of uterine fibroids who are initiating treatment with ESMYA.

Exclusion Criteria:

* Patient is pregnant or plans to become pregnant in the next 3 months,
* Patient is breastfeeding,
* Patient has genital bleeding of unknown etiology or not due to uterine fibroids,
* Patient has been diagnosed with uterine, cervical, ovarian or breast cancer,
* Patient is using an investigational drug/therapy or has discontinued the use of an investigational drug/therapy within 30 days prior to study enrollment,
* Patient has hypersensitivity to the active substance of ESMYA or to one of its excipients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target study population will include women who have had a diagnosis of symptomatic uterine fibroids and are initiating preoperative treatment with ESMYA.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-04 (Actual); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Occurrence of SAEs, adverse events (AEs) considered to be related to ESMYA or AEs leading to ESMYA treatment discontinuation. | Patients will be followed from baseline up to 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Oliver, MD, Study Director — PregLem SA
Locations (75):
- Austria (2):
  - LKH Klagenfurt, Klagenfurt
  - Private practice, Sankt Pölten
- France (8):
  - CHU Pellegrin Gynécologie, Bordeaux
  - Hopital Bicetre, Le Kremlin-Bicètre
  - CHU La Conception, Marseille
  - CHU Hôpital Mère-enfant, Nantes
  - Tenon CHU Paris Est, Paris
  - CHUV Maison Blanche Institut, Reims
  - CHU Anne de Bretagne, Rennes
  - CHU Tours Gynécologie, Tours
- Germany (25):
  - Universitätsklinikum Aachen, Aachen
  - Klinik am Hofgarten, Bayreuth
  - Charite, Berlin
  - Private practice, Berlin
  - Medizinisches Zentrum Bonn Friedensplatz, Bonn
  - Private Practice, Bruchsal
  - Private practice, Cologne
  - Private Practice, Diepholz
  - Private practive, Dorsten
  - Private practice, Dortmund
  - Frauenklinik, Universitätsklinikum Erlangen, Erlangen
  - Klinikum Esslingen, Esslingen am Neckar
  - Universitäts Frauenklinik, Freiburg im Breisgau
  - Gynäkologische Praxis, Geseke
  - Hormonzentrum Altonaerstrasse, Hamburg
  - Gynaekologische Praxisklinik Harburger Ring, Harburg
  - Private practice, Hoyerswerda
  - Private practice, Ilsede
  - Private practice, Krefeld
  - Gynäkologische Praxis, Mainz
  - Endoskopie und Endometriose Zentrum, München
  - Klinikum der Universitaet Muenchen - Klinik und Poliklinik für Frauenheilkunde, München
  - Private practice, Rodgau
  - Fachaerzte fuer Frauenheilkunde und Geburtshilfe, Rotenburg (Wümme)
  - Private practice, Völklingen
- Hungary (2):
  - Semmelweis University Faculty of Medicine, Budapest
  - University of Pécs Medical school, Pécs
- Italy (9):
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico S Orsola-Malpighi, Bologna
  - Universita di Cagliari, Cagliari
  - Azienda Ospedaliera Garibaldi-Nesima, Catania
  - Azienda Ospedaliera-universitaria di Ferrar-Arcispedale Sant'Anna, Cona
  - Università degli Studi di Firenze, Florence
  - Clinica ospedale san martino e cliniche universitarie convenzionate di genova, Genova
  - IRCCS ospedale maggiore policlinico mangiagalli e regina elena di milano, Milan
  - La Sapienza University, Roma
  - Ospedale Mauriziano "Umberto I", Torino
- Poland (7):
  - Private practice, Kętrzyn
  - Private practice, Komorów
  - Private practice, Lublin
  - Private Practice, Opole
  - Gravida Specjalistyczny Osrodek Ginekologii i Poloznictwa, Płock
  - Centrum Zdrowia mama i Ja, Wroclaw
  - Gabinet Ginekologiczny, Żory
- Portugal (2):
  - Hospital do Espirito santo de Évora, Evora
  - Hospital da Luz-Lisboa, Lisbon
- Romania (3):
  - Spitalul Clinic de Urgenta Militar Central, Bucharest
  - OG Clinic II " Dominic Stanca ", Cluj-Napoca
  - Spitalul Clinic de Urgenta, Târgu Mureş
- Spain (5):
  - Hospital del Mar, Barcelona
  - Hospital Sant Pau, Barcelona
  - Hospital de la Zarzuela, Madrid
  - Hospital Virgen de la Macarena, Seville
  - Hospital Virgen de la Salud, Toledo
- United Kingdom (12):
  - Bradford Royal Infirmary, Bradford
  - North Cumbria University Hospitals NHS Trust, Carlisle
  - Hull and East Yorshire Eye Hospital, East Yorkshire
  - Epsom & St Helier University Hospitals NHS Trust, Epsom Surrey
  - Royal devon and Exeter hospital, Exeter
  - Royal Hampshire County Hospital, Hampshire
  - University Hospitals of Leicester NHS Trust, Leicester
  - Liverpool Womens hospital, Liverpool
  - Barts and The London School of Medicine, London
  - King's College Hospital NHS Foundation, London
  - Nottingham University Hospital NHS trust, Nottingham
  - Southampton University Hospital, Southampton

REFERENCES:
- [Derived] Fernandez H, Descamps P, Koskas M, Lopes P, Brun JL, Darai E, Agostini A. Real-world data of 197 patients treated with ulipristal acetate for uterine fibroids: PREMYA study French population main outcomes. J Gynecol Obstet Hum Reprod. 2017 Sep;46(7):559-564. doi: 10.1016/j.jogoh.2017.06.006. Epub 2017 Jul 1. PMID 28676450